CLINICAL TRIAL: NCT01455870
Title: A Phase 3, Randomized, Active Comparator, Double-Blind, Multi-Center Study to Compare the Efficacy, Safety and Tolerability of ITCA 650 to Sitagliptin as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Brief Title: A Study to Evaluate ITCA 650 Compared to Sitagliptin as add-on Therapy for the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-105
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ITCA 650 60 mcg/day (Experimental): ITCA 650 is exenatide in DUROS
  Interventions: Drug: ITCA 650 60 mcg/day
- sitagliptin (Active Comparator): sitagliptin 100 mg/day
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: ITCA 650 60 mcg/day — exenatide in DUROS
  Arms: ITCA 650 60 mcg/day
Drug: sitagliptin — oral sitagliptin 100 mg/day
  Arms: sitagliptin

SUMMARY:
Phase 3 study to compare treatment with ITCA 650 to sitagliptin when added to metformin monotherapy in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 7.5% - 10.5%
* on metformin monotherapy
* BMI between 25 & 45 kg/m2

Exclusion Criteria:

* taking thiazolidinedione, sulfonylurea, DPP-4, exenatide, alpha glucosidase inhibitors, meglitinides or insulin within last 3 months
* history of pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c between Week 52 and Day 0 | 52 weeks

CONTACTS AND LOCATIONS:
Locations (51):
- United States (47):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Mateo, California
  - Tustin, California
  - Valley Village, California
  - Walnut Creek, California
  - Boca Raton, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Pembroke Pines, Florida
  - Canton, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - Franklin, Indiana
  - Greenfield, Indiana
  - Muncie, Indiana
  - Valparaiso, Indiana
  - Wichita, Kansas
  - Metairie, Louisiana
  - Brockton, Massachusetts
  - Traverse City, Michigan
  - Troy, Michigan
  - St Louis, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Endwell, New York
  - Morehead City, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Norman, Oklahoma
  - Bend, Oregon
  - Uniontown, Pennsylvania
  - Memphis, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tomball, Texas
- Rijeka, Croatia
- Hvidovre, Denmark
- Bad Lauterberg im Harz, Lower Saxony, Germany
- Riga, Latvia